CLINICAL TRIAL: NCT04670133
Title: Intervention With Inulin to Further Support Effectiveness of Sanative Therapy: Study Protocol for a Randomized Controlled Trial
Brief Title: Inulin Supplementation During Sanative Therapy to Further Improve Periodontal Healing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was planned before the COVID-19 pandemic and will not be pursued due to a change in research focus post-pandemic.
Sponsor: Brock University (Other)
Collaborators: Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-202
Record Dates: First submitted 2020-12-02; First posted 2020-12-17 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Periodontitis; Periodontal Diseases; Periodontal Pocket
Keywords: Sanative therapy; Scaling and root planing
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Periodontal Pocket | interventions — Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive one of the two treatments. They will be required to take one sachet per day (half in the morning; half in the evening) of the assigned intervention beginning 4 weeks before their scheduled sanative therapy appointment and remain on the intervention until 10 weeks after their sanative therapy appointment.
Who Masked: Participant, Care Provider
Masking Description: The intervention packages will be labelled with a unique code and there will be enough packages to account for the required number of participants. A member of the research team, not involved in providing the treatment, will be responsible for the randomization and labeling of the intervention packages, as well as creating a master list by matching the unique code to the treatment arm. The patient and care provider will be masked to the treatment arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inulin (Experimental): Supplementation with inulin for 4 weeks prior to and 10 weeks after sanative therapy. 10 g daily, divided into two equal doses.
  Interventions: Dietary Supplement: Inulin
- Placebo (Placebo Comparator): Supplementation with maltodextrin (as placebo) for 4 weeks prior to and 10 weeks after sanative therapy. 10 g daily, divided into two equal doses.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Inulin — Supplementation with a prebiotic, specifically inulin.
  Arms: Inulin
Dietary Supplement: Maltodextrin — Supplementation with maltodextrin (placebo)
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effectiveness of daily supplementation with inulin before, during and after sanative therapy (ST), on clinical outcomes of periodontal disease. The study design will allow the investigators to conclude if supplementation with inulin can favourably modulate oral microbiota prior to ST and can result in better periodontal health after ST.

DETAILED DESCRIPTION:
Periodontal disease is a chronic state of inflammation that can destroy the supporting tissues around the teeth, leading to a loss of connective tissue and the periodontal ligament, the resorption of alveolar bone and eventual tooth loss. Periodontal disease can also induce dysbiosis in the gut microbiome and contribute to low grade systemic inflammation. Prebiotic fibres such as inulin can selectively alter the intestinal microbiota to bring back a state of homeostasis by improving gut barrier functions and preventing inflammation. Through this mechanism, supplementation with inulin may be able to indirectly benefit periodontal health. The primary objective of this trial to determine if inulin supplementation, provided pre-sanative therapy (ST) through the healing phase (post-ST) is more effective than the placebo at improving clinical outcomes of periodontal health: decreasing both the number of sites with probing depths greater than or equal to 4 mm and increasing the absence of bleeding on probing (BOP). Secondary objectives include determining the effects of inulin supplementation pre- and post-ST on salivary markers of inflammation and periodontal-associated pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females age 19 years or older who are undergoing sanative therapy for moderate to severe chronic periodontitis are eligible
* Provided informed, written consent

Exclusion Criteria:

* Patients with severe periodontal disease that requires antibiotics with ST as part of their treatment
* Hemoglobin A1c levels greater than 8% in the previous 3 months
* Chronic GI conditions and/or infections (e.g. colon cancer, crohn's disease, inflammatory bowel disease, celiac disease and ulcerative colitis)
* Current or previous use of antibiotics for management of non-periodontal conditions within the past 3 month
* Current use of laxatives, prebiotics, probiotics and/or fibre supplements
* Smokers and/or cannabis users
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Probing depth | At pre-sanative therapy
  This is a routine clinical measure of periodontal health (measured in mm)
Probing depth | At post-sanative therapy (10 weeks after sanative therapy is completed)
  This is a routine clinical measure of periodontal health (measured in mm)
Bleeding on probing (BOP) | At pre-sanative therapy
  This is a clinical measure of inflammation and represented as the percentage to bleeding sites that are measured at 6 sites per tooth
Bleeding on probing (BOP) | At post-sanative therapy (10 weeks after sanative therapy is completed)
  This is a clinical measure of inflammation and represented as the percentage to bleeding sites that are measured at 6 sites per tooth

SECONDARY OUTCOMES:
Salivary markers of inflammation | At pre-sanative therapy
  Levels of interleukin (IL)-1beta, IL-6, C-reactive protein (CRP), Matrix metalloproteinase-8 will be measured.
Salivary markers of inflammation | At sanative therapy (6 weeks after pre-sanative appointment)
  Levels of interleukin (IL)-1beta, IL-6, C-reactive protein (CRP), Matrix metalloproteinase-8 will be measured.
Salivary markers of inflammation | At post-sanative therapy (10 weeks after sanative therapy is completed)
  Levels of interleukin (IL)-1beta, IL-6, C-reactive protein (CRP), Matrix metalloproteinase-8 will be measured.
Periodontal-Associated Pathogens | At pre-sanative therapy
  Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola will be measured by quantitative polymerase chain reaction (PCR).
Periodontal-Associated Pathogens | At sanative therapy (6 weeks after pre-sanative appointment)
  Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola will be measured by quantitative PCR.
Periodontal-Associated Pathogens | At post-sanative therapy (10 weeks after sanative therapy is completed)
  Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola will be measured by quantitative PCR.
Dietary assessment | At pre-sanative therapy
  Intake of energy, carbohydrate, fat and protein will be measured with the automated self-administered dietary intake (ASA-24) questionnaire. This is an online food recall that patients will complete three times for each visit, reporting on their dietary intake from the last 24 hours.
Dietary assessment | At sanative therapy (6 weeks after pre-sanative appointment)
  Intake of energy, carbohydrate, fat and protein will be measured with the automated self-administered dietary intake (ASA-24) questionnaire. This is an online food recall that patients will complete three times for each visit, reporting on their dietary intake from the last 24 hours.
Dietary assessment | At post-sanative therapy (10 weeks after sanative therapy is completed)
  Intake of energy, carbohydrate, fat and protein will be measured with the automated self-administered dietary intake (ASA-24) questionnaire. This is an online food recall that patients will complete three times for each visit, reporting on their dietary intake from the last 24 hours.
Body Mass Index | At pre-sanative therapy
  Body weight and height will be measured to calculate BMI
Body Mass Index | At sanative therapy (6 weeks after pre-sanative appointment)
  Body weight and height will be measured to calculate BMI
Body Mass Index | At post-sanative therapy (10 weeks after sanative therapy is completed)
  Body weight and height will be measured to calculate BMI

CONTACTS AND LOCATIONS:
Overall Officials: Wendy E Ward, PhD, Principal Investigator — Brock University

REFERENCES:
- [Derived] Zanatta CAR, Fritz PC, Comelli EM, Ward WE. Intervention with inulin prior to and during sanative therapy to further support periodontal health: study protocol for a randomized controlled trial. Trials. 2021 Aug 10;22(1):527. doi: 10.1186/s13063-021-05504-1. PMID 34376241